CLINICAL TRIAL: NCT07165847
Title: Neoadjuvant Radiotherapy Plus Tegafur, Oxaliplatin and Iparomlimab and Tuvonralimab in Resectable Gastric and GE-junction Cancer : A Randomized, Two-arm, Prospective Trial (TRIUNITE-05)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025 (64-01)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Immunotherapy; Gastric Cancer (GC); Radiotherapy; Neoadjuvant Therapy; Neoadjuvant Chemoimmunotherapy
Keywords: Immunotherapy; Gastric Cancer; Radiotherapy; Neoadjuvant therapy; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Tegafur; Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Stage 1: Radiotherapy (30 Gy/10 fractions) Stage 2: 6 cycles immunochemotherapy(SOX + Iparomlimab and Tuvonralimab (5 mg/kg, i.v.))
  Interventions: Drug: Iparomlimab and Tuvonralimab; Drug: Oxaliplatin; Drug: Tegafur; Radiation: Radiotherapy
- Group B (Experimental): Stage 1: 3 cycles immunochemotherapy (SOX + Iparomlimab and Tuvonralimab (5 mg/kg, i.v.)) Stage 2: Radiotherapy (30 Gy/10 fractions) Stage 3: 6 cycles immunochemotherapy (SOX + Iparomlimab and Tuvonralimab (5 mg/kg, i.v.))
  Interventions: Drug: Iparomlimab and Tuvonralimab; Drug: Oxaliplatin; Drug: Tegafur; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — q3w Iparomlimab and Tuvonralimab 5mg/kg on day 1 of each cycle
Drug: Oxaliplatin — 130mg/m2 on day 1 of each cycle
Drug: Tegafur — <1.25 m2, 40 mg; 1.25 to ≤1.5 m2, 50 mg; and ≥ 1.5 m2, 60 mg；po；d1-14 bid
Radiation: Radiotherapy — 30 Gy/10 fractions

SUMMARY:
Neoadjuvant radiotherapy plus Tegafur, Oxaliplatin and Iparomlimab and Tuvonralimab in Resectable Gastric and GE-junction Cancer : A Randomized, Two-arm, Prospective Trial (TRIUNITE-05)

DETAILED DESCRIPTION:
TRIUNITE-05 is a randomized, two-arm, uncontrolled, prospective study to evaluate the efficacy and safety of neoadjuvant radiotherapy combined with immunochemotherapy for locally advanced G/GEJ adenocarcinoma. This study will include subjects with locally progressive G/GEJ adenocarcinoma, patients in Group A will be treated with radiotherapy (30Gy/10f) followed by sequential SOX regimen in combination with Iparomlimab and Tuvonralimab (5 mg/kg, i.v.) for 6 cycles of induction therapy, with full evaluation and surgery 4-6 weeks after the end of the treatment; patients in group B will be treated with SOX regimen in combination with Iparomlimab and Tuvonralimab for 3 cycles of induction therapy followed by sequential radiotherapy ( 30Gy/10f) followed by 3 cycles of sequential SOX regimen combined with Iparomlimab and Tuvonralimab (5 mg/kg, i.v.), with full evaluation and surgery 4~6 weeks after the end of treatment. For those who were assessed to be inoperable after neoadjuvant therapy, the original regimen of immunotherapy in combination with chemotherapy was concurrently administered until progression; if it was ineffective, the regimen was changed to a second-line chemotherapy regimen or other anti-tumor combination therapy regimens were considered as appropriate. Patients were then entered into long-term survival follow-up. During the study period, preoperative and postoperative blood, feces, and pathological tissues of subjects were collected for testing biomarkers to explore the potential benefit population of neoadjuvant therapy. Blood and fresh tissues were subjected to single-cell sequencing, spatial transcriptomic or proteomic analysis, and tissues were subjected to multiplex immunofluorescence assay, in order to further search for potential biomarkers that may be beneficial for the benefit of neoadjuvant therapy in locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patients are able to understand and voluntarily sign the written informed consent, which must be signed prior to the implementation of the designated research procedures required by the study.
* The age at the time of signing the informed consent form (ICF) is ≥ 18 years old, both male and female.
* Histologically confirmed to have HER2-negative gastric or gastroesophageal junction adenocarcinoma (Siewert type II or Siewert type III with ≤2 cm of esophageal involvement) with AJCC 8th edition staging of Stage IIA- Stage III, i.e., T1- 2N+, and T3-4 and or N+, and resectable;.
* The patients are willing to provide fresh blood, feces, and tumor tissue for biomarker analysis, and the tissue samples provided are of sufficient quality to evaluate the status of biomarkers. If sufficient tissue is not provided, repeated sampling may be required.
* The patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
* The expected survival time was ≥ 3 months.\
* No previous anti-tumor therapy (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy, and traditional Chinese medicine with clear anti-tumor effects, excluding abdominal exploration for diagnostic staging);
* The patient has adequate organs function

  1. The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1.5*10^9/L, hemoglobin ≥90g/L (5.58 mmol/L), and platelets ≥100*10^9/L.
  2. The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥50 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed).
  3. The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 μmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).
  4. The patient must have adequate coagulation function as defined by international normalized ratio (INR) ≤1.5
* Within 7 days before the first administration, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraceptives during the study period and within 180 days after the last administration. In this program, women of childbearing age are defined as sexually mature women:

  1. No hysterectomy or bilateral ovariectomy
  2. Natural menopause does not last for 24 months (amenorrhea after cancer treatment does not rule out fertility) (that is, menstruation occurs at any time in the previous 24 months).

For male patients whose sexual partners are women of childbearing age, they must agree to use effective contraception during the study drug use and within 180 days after the last administration.

Exclusion Criteria:

* Palliative local treatment was given to non-target lesions within 2 weeks before the first administration, and systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) was received within 2 weeks before the first administration. Chinese herbal medicine or proprietary Chinese medicine with anti-tumor indications was received within 2 weeks before the first administration.
* The patient has previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy, etc. any treatment aimed at the immune mechanism of tumor.
* There was a history of gastrointestinal perforation and gastrointestinal fistula within 6 months before the first administration. If the perforation or fistula has been removed or repaired, and the disease has been judged by the researchers to recover or remission, it may be allowed to join the group.
* Active or previously recorded inflammatory bowel disease (such as Crohn's disease or ulcerative colitis). Unable to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal diseases that seriously affect drug use and absorption.
* There were active malignant tumors in the past 3 years, except for tumors that participated in the study and local tumors that had been cured. such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast cancer in situ, localized prostate cancer and so on.
* Active or untreated brain metastases, meningeal metastases, spinal cord compression or leptomeningeal diseases are known.

However, the patients who met the following requirements and had measurable lesions outside the central nervous system were allowed to enter the group: asymptomatic after treatment, imaging was stable for at least 4 weeks before the start of treatment (such as no new or enlarged brain metastases). And systemic corticosteroids and anticonvulsant drugs have been stopped for at least 2 weeks.

* There are pleural effusion with clinical symptoms, pericardial effusion or ascites requiring frequent drainage (≥ 1 / month).
* Study active autoimmune diseases that require systematic treatment within 2 years before the start of treatment, or researchers determine the existence of autoimmune diseases that may recur or plan treatment. Except for the following:

  1. Skin diseases that do not require systematic treatment (e.g. vitiligo, hair loss, psoriasis or eczema)
  2. Hypothyroidism caused by autoimmune thyroiditis requires only a stable dose of hormone replacement therapy.
  3. Type I diabetes mellitus requiring only a stable dose of insulin replacement therapy
  4. Asthma has been completely relieved in childhood and no intervention is needed in adults.
  5. The researchers determined that the disease would not recur without external triggers.
* There are any of the following cardio-cerebrovascular diseases or cardio-cerebrovascular risk factors:

  1. Within 6 months before the first administration, there were myocardial infarction, unstable angina pectoris, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (according to New York Heart Association functional grade 2 or above), symptomatic or poorly controlled arrhythmia, or any arterial thromboembolic event.
  2. There was a history of deep venous thrombosis, pulmonary embolism or other severe thromboembolism within 3 months before the first administration.
  3. There are major vascular diseases, such as aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis, which may be life-threatening or require surgery within 6 months.
  4. Previous history of myocarditis and cardiomyopathy.
  5. Left ventricular ejection fraction (LVEF) < 50%.
* Toxicity that has not been alleviated by previous antineoplastic therapy is defined as undiminished to Grade 0 or 1 of the National Cancer Institute (NCI) General terminology Standard for adverse events (CTCAE) (NCICTCAEv5.0), or to the level specified in the selection / exclusion criteria, with the exception of alopecia / pigmentation. The patients who develop irreversible toxicity and are not expected to increase after drug administration (such as hearing loss) may be included in the study after consultation with researchers. Long-term toxicity caused by radiotherapy may be included in the study after consultation with the researchers who are determined by the researchers to be unable to recover.
* Grade 2 peripheral nerve disease was defined according to NCI CTCAE v5.0 standard.
* Interstitial lung disease or non-infectious pneumonia is known to be symptomatic or requires systemic glucocorticoid treatment in the past, and researchers have determined that it may affect toxicity assessment or management associated with research treatment.
* Active tuberculosis is known to exist. The patients suspected of having active pulmonary tuberculosis should be examined for chest X-ray, sputum and excluded by clinical symptoms and signs.
* Received systemic anti-infective therapy (excluding antiviral therapy for hepatitis B or C) within 2 weeks before the first administration.
* The history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation are known.
* There are clinical active hemoptysis, active diverticulitis, abdominal abscess and gastrointestinal obstruction.
* There were significant clinical bleeding symptoms or definite bleeding tendency within 1 month before the first administration, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis.
* It is known that endoscopy shows signs of active bleeding.
* There were other major operations in addition to the diagnosis of gastric cancer within 28 days before the first administration.
* Untreated active hepatitis B patients (HBsAg positive and HBV-DNA more than 1000 copies / ml [200IU/ml] or higher than the detection lower limit), patients with hepatitis B were required to receive anti-HBV treatment during the study treatment; active hepatitis C patients (HCV antibody positive and HCV-RNA levels higher than the detection lower limit).
* Those who are known to have a history of immunodeficiency or are HIV positive.
* Known active syphilis infection.
* Is participating in another clinical study, unless it is a follow-up period for observational, non-interventional clinical studies or interventional studies.
* The patients who needed systemic treatment with glucocorticoids (> 10mg/ prednisone or equivalent dose) or other immunosuppressive drugs within 14 days before the first administration. Except for the following:

  1. If there is no active autoimmune disease, inhaled, ophthalmic or topical glucocorticoids or doses of ≤ 10mg/ prednisone or equivalent doses of other glucocorticoids are allowed.
  2. Physiological dose of systemic glucocorticoid ≤ 10mg/ prednisone or equivalent dose of other glucocorticoids.
  3. Glucocorticoids are used as pretreatment of infusion-related reactions or allergic reactions (such as medication before CT examination).
* The live vaccine was given within 30 days of the first administration, or is planned during the study period.
* A history of severe hypersensitivity to other monoclonal antibodies is known.
* It is known to be unable to meet the requirements of the trial because of mental illness or substance abuse disorder.
* The patients who are known to have a history of allergy or hypersensitivity to drugs or any of its components in the combined immunotherapy regimen.
* The patient is pregnant or breastfeeding.
* The researchers believe that there may be a risk of receiving the study drug treatment, or any condition that will interfere with the evaluation of the study drug or the safety of the patients or the interpretation of the research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2028-09-23 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 8 months

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) | 8 months
Objective Response Rate (ORR) | 7 months
Disease Control Rate (DCR) | 7 months
Progression Free Survival (PFS) | 3 years
Overall Survival (OS) | 3 years
Clinical Complete Response (cCR) | 7 months

OTHER OUTCOMES:
Adverse events (AE) | 6 months
Correlation analysis of evaluating the relationship between clinicopathological characteristics and neoadjuvant immunochemotherapy and radiotherapy | 3 years
Correlation analysis of evaluating the relationship between multi-omics analysis of tumor tissue and neoadjuvant immunochemotherapy efficacy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Principal Investigator — Army Medical Center of the People's Liberation Army
Locations (1):
- Army Medical Center, Chongqing, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: Undecided